CLINICAL TRIAL: NCT04101123
Title: Social Inequalities in the Participation and Activity in Children and Adolescents With Leukemia, Brain Tumors, and Sarcomas
Brief Title: Children and Adolescents With Leukemia, Brain Tumors, and Sarcomas
Acronym: SUPATEEN
Status: Completed | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Julia Roick, Research Associate, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: 70113424
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Leukemia; Brain Tumor; Sarcoma; Childhood Cancer; Cancer; Adolescent Cancer
Keywords: Social inequalities; Social dimensions of health; Brain tumors; Leukemia; Sarcomas; Childhood Cancer; Children and adolescents with cancer
MeSH Terms: conditions — Leukemia; Brain Neoplasms; Sarcoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adolescents with cancer: Children and adolescents between 10-18 years with newly diagnosed leukemia, brain tumors, and sarcomas
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
Aim of this study is to investigate the influence of social factors on participation and activity among children and adolescents aged 10-18 years with leukemia, brain tumors, and sarcomas. Furthermore personal and treatment-related factors and their impact on participation will be explored

DETAILED DESCRIPTION:
Background: About 2000 children and adolescents under the age of 18 develop cancer each year in Germany. Because of more differentiated diagnostics and standardized treatment protocols, a high survival rate can be reached for many types of the disease. Nevertheless, patients face a number of long-term effects related to the treatment. As a result, physical and psychological consequences have increasingly become the focus of research in recent years. Social dimensions of health have rarely been investigated in pediatric oncology so far. Yet, there are no robust results that allow an estimation of whether and to what extent the disease and treatment impair the participation of children and adolescents and which factors mediate this effect. Social participation is of great importance especially because interactions with peers and experiences in different areas of life are essential for the development of children and adolescents.

Methods: Data are collected in a longitudinal, prospective, observational multicenter study. For this purpose, all patients and their parents who are being treated for cancer in one of the participating clinics throughout Germany will be interviewed within the first month after diagnosis (t1), after completion of intensive treatment (t2) and half a year after the end of intensive treatment (t3) using standardized questionnaires. Analysis will be done by descriptive and multivariate methods.

Recruitment: Patients will be consecutively recruited in one of the participating clinics throughout Germany.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed with confirmed leukemia, brain tumor or sarcoma
* age 10-18 years
* written informed consent of the patient and of one of the parents if they are under the age of 18

Exclusion Criteria:

* having a relapse or secondary tumor
* insufficient command of German
* profound cognitive and physical impairments

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with leukemia, brain tumors, and sarcomas who are between 10 to 18 years old and their parents
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Social participation and activity | Within the first month after diagnosis until half a year after intensive treatment
  The Child and Adolescent Scale of Participation, CASP
Level of quality of life | Within the first month after diagnosis until half a year after intensive treatment
  Questionnaire to assess Health Related Quality of Life in chronically ill Children and Adolescents, KINDL Subscales: physical well-being, emotional well-being, self-esteem, family, friends, school, and a total score Values: range from 0 to 100 (higher values represent better quality of life)

SECONDARY OUTCOMES:
Evaluation of the treatment | End of intensive treatment
  Questionnaire to assess the Satisfaction with the Treatment, FBB Subscales: success of treatment (range 0-20), relationship to medical team (range 0-28), treatment conditions (range 0-24), and a total score (range 0-72) Values: higher values represent better evaluation
Self-concept | Within the first month after diagnosis until half a year after intensive treatment
  Self-Description Questionnaire, SDQ
Fatigue | Within the first month after diagnosis until half a year after intensive treatment
  Subscale Fatigue from the Questionnaire to assess Quality of Life of Cancer Patients developed by the European Organisation for Research and Treatment of Cancer, EORTC QLQ-C30 Values: range from 0 to 100 (higher values represent higher symptoms of fatigue)
Social support | Within the first month after diagnosis until half a year after intensive treatment
  Social Support Scale, SSS Values: total score with a range 8-40 (higher values represent higher support)
Illness perception | Within the first month after diagnosis until half a year after intensive treatment
  Illness Perception Questionnaire, IPQ
Self-efficacy | Within the first month after diagnosis until half a year after intensive treatment
  General Self-Efficacy Scale; SWE
Optimism | Within the first month after diagnosis until half a year after intensive treatment
  Subscale from The Bern Subjective Well-Being Questionnaire for Adolescents, BFW
Psychosocial problems and strengths | Within the first month after diagnosis until half a year after intensive treatment
  Strengths and Difficulties Questionnaire, SDQ Subscales: emotional problems, conduct problems, peer problems, hyperactivity, and prosocial behavior Values: each scale has a range 0-10 (higher values represent higher problems except prosocial behavior)
Sense of coherence | Within the first month after diagnosis until half a year after intensive treatment
  Children Sense of Coherence Scale, C-SOC
Coping | Within the first month after diagnosis until half a year after intensive treatment
  Coping Questionnaire for Children and Adolescents, CODI
Mental health | Within the first month after diagnosis until half a year after intensive treatment
  Children's Depression Screener, Child-S
Autonomy | Within the first month after diagnosis until half a year after intensive treatment
  Subscale from The Kidscreen Questionnaire

OTHER OUTCOMES:
Parental coping with chronic childhood disease | Within the first month after diagnosis until half a year after intensive treatment
  Coping Health Inventory for Parents, CHIP (parental questionnaire)
Psychosocial needs | Within the first month after diagnosis until the end of intensive treatment
  Short-Form Supportive Care Needs Survey Questionnaire, SCNS-SF34 (parental questionnaire)
Evaluation of the treatment | End of intensive treatment
  Questionnaire to assess the Satisfaction with the Treatment, FBB
Familial burden | End of intensive treatment until half a year after intensive treatment
  Impact on Family Scale in Families with Children with Disabilities, FaBel (parental questionnaire)
Family resources | Within the first month after diagnosis and half a year after intensive treatment
  Family Environment Scale, FES (parental questionnaire)
Satisfaction with life | Within the first month after diagnosis until half a year after intensive treatment
  The Satisfaction With Life Scale, SWL
Doctor-parent relationship | End of intensive treatment
  Patient Reactions Assessment, PRA-D
Level of quality of life | Within the first month after diagnosis until half a year after intensive treatment
  The Short Form Health Survey, SF-12
Sense of coherence | Within the first month after diagnosis until half a year after intensive treatment
  Sense of Coherence Scale - Leipziger Short Form, SOC-L9
Mental health | Within the first month after diagnosis until half a year after intensive treatment
  Hospital Anxiety and Depression Scale, HADS

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Richter, Prof. Dr., Study Chair — Martin-Luther-Universität Halle-Wittenberg
Locations (1):
- Institute of Medical Sociology, Halle, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roick J, Berner R, Bernig T, Erdlenbruch B, Escherich G, Faber J, Klein C, Bochennek K, Kratz C, Kuhr J, Langler A, Lode HN, Metzler M, Muller H, Reinhardt D, Sauerbrey A, Schepper F, Scheurlen W, Schneider D, Schwabe GC, Richter M. Social inequalities in the participation and activity of children and adolescents with leukemia, brain tumors, and sarcomas (SUPATEEN): a protocol for a multicenter longitudinal prospective observational study. BMC Pediatr. 2020 Jan 31;20(1):48. doi: 10.1186/s12887-020-1943-3. PMID 32005112